CLINICAL TRIAL: NCT01973842
Title: Evaluation of the Optimal Dose of GnRH Agonist for Triggering Final Oocyte Maturation in High Risk OHSS Patients Undergoing Ovarian Stimulation for IVF With GnRH Antagonists and Recombinant FSH.
Brief Title: Evaluation of the Optimal Dose of GnRH Agonist for Triggering Final Oocyte Maturation in High Risk OHSS Patients
Acronym: ATD
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aristotle University Of Thessaloniki (Other)
Collaborators: Eugonia IVF Unit, Athens, Greece (Other)
Responsible Party: Principal Investigator, E.M. Kolibianakis, Ass Professor in Obstetrics - Gynecology and Assisted Reproduction, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Agonist triggering dose
Record Dates: First submitted 2013-10-25; First posted 2013-11-01 (Estimated); Last update posted 2016-02-12 (Estimated); Status verified 2016-02

CONDITIONS: Subfertility
Keywords: GnRH agonist; OHSS; Triggering final oocyte maturation
MeSH Terms: conditions — Infertility | interventions — Triptorelin Pamoate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 0.2 mg triptorelin (Active Comparator): 0.2 mg triptorelin compared with 0.1 mg triptorelin and 0.4 mg triptorelin
  Interventions: Drug: 0.2 mg triptorelin
- 0.1 mg triptorelin (Active Comparator): 0.1 mg triptorelin compared with 0.2 mg triptorelin and 0.4 mg triptorelin
  Interventions: Drug: 0.1 mg triptorelin
- 0.4 mg triptorelin (Active Comparator): 0.4 mg triptorelin compared with 0.1 mg triptorelin and 0.2 mg triptorelin
  Interventions: Drug: 0.4 mg triptorelin

INTERVENTIONS:
Drug: 0.1 mg triptorelin
  Arms: 0.1 mg triptorelin
Drug: 0.2 mg triptorelin
  Arms: 0.2 mg triptorelin
Drug: 0.4 mg triptorelin
  Arms: 0.4 mg triptorelin

SUMMARY:
The present study aims to investigate whether the dosage of the GnRH agonist used for triggering final oocyte maturation affects the maturity of the oocytes retrieved in high risk for OHSS patients undergoing ovarian stimulation for IVF using GnRH antagonists and recombinant FSH.

DETAILED DESCRIPTION:
Three different doses of GnRH agonist (0.1mg, 0.2mg or 0.4 mg) will be used randomly to trigger final oocyte maturation. The primary outcome measure will be the percentage of mature oocytes retrieved.

Secondary outcomes will include: number of oocytes retrieved, oocyte recovery rate (number of oocytes retrieved/ number of follicles >11mm in diameter on the day of triggering), fertilization rates and OHSS occurrence.

Serum LH, FSH, E2, PRG levels will be assessed at 8-36 hours following agonist administration and on days 3-4-7-10 after triggering final oocyte maturation.

ELIGIBILITY:
Inclusion Criteria: Patients undergoing ovarian stimulation for IVF using GnRH antagonist protocol

* Age < 40 years
* Anticipated high ovarian response

Exclusion Criteria:

* Endometriosis > than grade II
* One ovary

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2014-02; Primary Completion 2016-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Percentage of mature oocytes retrieved | 36 hours post GnRH agonst administration
  Percentage of mature oocytes retrieved following oocyte retrieval

SECONDARY OUTCOMES:
total number of oocytes retrieved | 36 hours post GnRH agonist administration
oocyte recovery rate | 36 hours post GnRH agonist administration
Fertilization rate | Day 1 post oocyte retrieval
Serum LH, FSH, E2, PRG levels | 8-36 hours post triggering and on days 3-4-7-10 after GnRH agonist administration
Duration of luteal phase | 16 days
OHSS occurrence | 16 days post triggering
  Occurrence of ovarian hyperstimulation syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Efstratios Kolibianakis, MD, MSc, PhD, Principal Investigator — Unit of Human Reproduction, 1st Dept of Obstetrics and Gynaecology, Medical School, Aristotle University of Thessaloniki Thessaloniki, Greece
Locations (2):
- Greece (2):
  - Eugonia IVF Unit, Athens
  - Unit of Human Reproduction, 1st Dept of Obstetrics and Gynaecology, Medical School, Aristotle University of Thessaloniki, Thessaloniki